CLINICAL TRIAL: NCT05691179
Title: The Association of COVID-19 Infection and Relapse of Idiopathic Membranous Nephropathy
Brief Title: COVID-19 Infection and Idiopathic Membranous Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Pinggu District Hospital (Other); Beijing Fangshan District Liangxiang Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Professor Wenhu Liu, Beijing Friendship Hospital
Other Study IDs: 2022-P2-429-01
Record Dates: First submitted 2023-01-18; First posted 2023-01-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infection group: the patients with IMN and COVID-19 infection

SUMMARY:
Infection is one of common risk factors for relapsing of idiopathic membranous nephropathy (IMN). However, it is still unclear wheather COVID-19 infection can induce the relapsing of IMN. Herein, in this prospective, multi-center, cohort study, the investigator enrolled the IMN patients with COVID-19 infection.

All subjects will be followed for three months with four visits at 1, 2 and 3 months. Then the investigator will compare the rate of replase of IMN in the two groups to evaluate the association of COVID-19 infection and replapse of IMN.

ELIGIBILITY:
Inclusion Criteria:

1. the status of nephrotic syndrome is complete remmision or partial remmision;
2. estimated glomerular filtration rate (eGFR according to the CKD-EPI formula) ≥60 mL/min per 1.73 m2;
3. patients with a moderate risk of IMN.

Exclusion Criteria:

1. secondary causes of MN;
2. the labarotary data two months before enrolement is absent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All eligible IMN patients with COVID-19 infection can be enrolled.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 3 months
  relaspe of nephrotic syndrome: proteinuria<0.3g/d, serum albumin>30g/l, serum creatitine below 111 μmol/l

SECONDARY OUTCOMES:
secondary outcome | 0.5, 1, and 2 months
  relaspe of nephrotic syndrome: proteinuria<3.5g/d (decreased over 50% of baseline), serum albumin>30g/l, steady serum creatitine (fluctuated less than 20% of baseline), meet the above criteria over 2 times

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Friedship Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Beijing Liangxiang Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No